CLINICAL TRIAL: NCT03383172
Title: Mental Health Prevention Among Preschool Children: a Pilot Study of the Adaptation of the I Can Problem Solve (ICPS) Program to Chile
Brief Title: Mental Health Prevention Among Preschool Children Using a Culturally Adapted Version of ICPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación San Carlos de Maipo (Other)
Collaborators: Universidad de los Andes, Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FSCM170505
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Mental Health; Aggressive Childhood Behavior; Problem Behavior; Social Behavior
Keywords: Prevention; Promotion; Mental Health
MeSH Terms: conditions — Psychological Well-Being; Problem Behavior; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ICPS with internal school facilitator (Experimental): Schools with preschool students. All consented students in the class will participate in the ICPS preschool program, adapted to the Chilean reality and culture. The program is manualized and will be delivered by the early educator of the class, who is part of the school personnel.This internal facilitator will be trained in the program. Each of the 59 sessions lasts around 20 minutes, delivered 2 to 3 times a week, during 5 months. ICPS content includes vocabulary and concepts about emotions, and the development of problem-solving skills, practising alternative solutions, consequences and the sequential thought (solutions-consequences). Interactive techniques (e.g. games, role-playing, and the use of stories, illustrations and puppets), and guided discussion strategies are used to solve problems.
  Interventions: Behavioral: I Can Problem Solve (ICPS) Program
- ICPS with external facilitator (Active Comparator): Schools with preschool students. All consented students in the class will participate in the ICPS preschool program, adapted to the Chilean reality and culture. The program is manualized and will be delivered by an external trained early educator, who is part of the research team. The early educator of the class, who is part of the school personnel, will also be trained to collaborate with all the program activities with the external facilitator. Each of the 59 sessions lasts around 20 minutes, delivered 2 to 3 times a week, during 5 months. ICPS content includes vocabulary and concepts about emotions, and the development of problem-solving skills, practising alternative solutions, consequences and the sequential thought (solutions-consequences). Interactive techniques (e.g. games, role-playing, and the use of stories, illustrations and puppets), and guided discussion strategies are used to solve problems.
  Interventions: Behavioral: I Can Problem Solve (ICPS) Program
- Control Group (No Intervention): School in the control group will continue to carry out their normal academic and prevention activities.

INTERVENTIONS:
Behavioral: I Can Problem Solve (ICPS) Program — The 59 sessions of ICPS program explicitly promote cognitive regulation, solving social problems, and emotional learning skills.
  Other Names: Interpersonal Cognitive Problem Solving Program
  Arms: ICPS with external facilitator; ICPS with internal school facilitator

SUMMARY:
Mental health in Chilean children and families is an urgent public health problem. Prevalence of psychiatric disorders among children between 4 and 11 years old is 27.8%, a higher percentage than was found in adolescents between 12 and 18 years old, which is 16.5%. The most frequent disorders in the population between 4 and 11 years old were disruptive disorders (20.6%), followed by anxiety disorders (9.2%). Mental health problems generate a high burden of disease on society in general; and there is an important treatment gap, especially among economically vulnerable populations. Prevention strategies appear to be the more recommendable options, mainly if these interventions can be implemented early in life and at low cost. Few preventive interventions aiming to increase resilience in the face of adversity, have been rigorously evaluated in Chile among preschoolers. There is substantial international evidence that shows that strengthening basic psychological skills, such as emotion regulation and social problem-solving, can reduce the incidence of mental pathology and improve various academic indicators. The curriculum of the Interpersonal Cognitive Problem Solving Program, also known as I Can Problem Solve (ICPS), is focused on the development of the cognitive process and children's social problem-solving skills. ICPS has been found to be effective in increasing pro-social behaviours and reducing aggressive behaviour among preschoolers. No previous studies in Spanish-speaking Latin American countries have been conducted aiming to explore the acceptability and feasibility of ICPS to provide information to evaluate later the effectiveness of this intervention at a larger scale.

The main objective of this study is the evaluation of the acceptability and feasibility of an adapted version of ICPS in the national context at educational institutions with high socio-economic vulnerability, with the ultimate goal of increasing social-emotional competence and reducing emotional and behavioural problems in preschoolers.

DETAILED DESCRIPTION:
Background. Mental health in Chilean children and families is an urgent public health problem. Several epidemiological studies have shown that a significant percentage of the adult population has psychiatric disorders. For example, one recent study showed that 31.5% of the population aged 15 and over has some type of psychiatric pathology in their lives, and that 22.2% suffered from a mental disorder during the last year (Vicente et al., 2006). Today we know that many of the disorders present in the adult population begin in childhood and adolescence and that preventing their onset can have a significant impact on the future functioning of the individual. The few epidemiological studies on the Chilean child and adolescent populations show that the prevalence of psychiatric disorders among children between 4 and 11 years old is 27.8%, a higher percentage than was found in adolescents between 12 and 18 years old, which is 16.5% (Vicente et al., 2012). The most frequent disorders in the population between 4 and 11 years old were disruptive disorders (20.6%), followed by anxiety disorders (9.2%) (Vicente et al., 2012). Mental health problems generate a high burden of disease on society in general (Patel, et al., 2016); and there is an important gap in the treatment of these, especially in populations that are more economically vulnerable (Patel, et al., 2016). Prevention strategies appear to be the more recommendable options, mainly if these interventions can be implemented early and at low cost. Few preventive interventions, or interventions that increase resilience in the face of adversity, have been rigorously evaluated in Chile. There is substantial evidence that shows that strengthening social and emotional learning skills can reduce the incidence of mental pathology and improve various academic indicators (Domitrovich et al., 2017). These social-emotional skills include the ability to identify and express emotions, to be able to adapt to social context, to regulate emotions, the ability to inhibit behaviour, and problem-solving skills (Denham, 2006; Domitrovich et al., 2017). Deficits in these skills have been associated with the appearance of both internalization problems (emotional problems such as depression and anxiety) and externalization problems (such as disruptive behavioural problems), as well as peer rejection (Garner & Waajid, 2012).

The curriculum of the Interpersonal Cognitive Problem Solving Program, also known as I Can Problem Solve (ICPS) (Shure, 1992), is focused on the development of the cognitive process and children's social problem-solving skills. That is, it is a program that explicitly promotes cognitive regulation (skills for listening and paying attention, sequencing and planning tasks) and solving social problems (thinking up alternative solutions, causal thinking, means-to-an-end thinking, and sequential planning). But it also includes the promotion and learning of emotional processes (particularly emotional expression/knowledge, perspective, and empathy) (Jones et al., 2017). Several studies conducted among disadvantaged population have shown that students who received ICPS had better results regarding increasing pro-social behaviours and reducing aggressive behaviour compared with students in the control group (Shure & Spivack, 1982; Boyle & Hassett-Walker, 2008). ICPS is a universal intervention designed to promote interpersonal cognitive processes and problem-solving skills in children from preschool through 6th grade. This project will adapt the preschool program, which has a total of 59 sessions. Each session lasts around 20 minutes, and the trained facilitator follows a simple manual that guides their work with the students on ICPS vocabulary and concepts and the development of problem-solving skills such as practising alternative solutions, consequences and the sequential thought (solutions-consequences). An interactive technique and guided discussion strategies are used to solve problems. Interactive methods include games, role-playing, and the use of stories, illustrations and puppets. These contents may also be used in other curricular activities for children, whether they are working on Math, Reading or Science. Children learn how to think and not what to think.

Aims. The general objective of this study is the evaluation of the acceptability and feasibility of an adapted version of ICPS in the national context at educational institutions with high socio-economic vulnerability, with the ultimate goal is of increasing social-emotional competence and reducing emotional and behavioural problems in preschoolers.

Methods. A pilot study consisting of two phases. Firstly, a formative stage when all intervention evaluation materials will be prepared, including the validation of instruments assessing socio-emotional skills; and curriculum of ICPS Preschool Program will be translated, edited and adapted, working closely with the author of the program Dr Myrna Shure. Secondly, the program will be implemented using a three-arm randomised controlled trial design. The acceptability and feasibility of its implementation in the national context will be evaluated, and changes in the development of social-emotional skills, behavioural problems and mental health, before and after the intervention. There will be two Intervention groups: 1) Schools implementing the ICPS program delivered by the school early teacher, trained by the research team; and 2) Schools implementing the ICPS program delivered by an early teacher hired and trained by the research team, who will work collaboratively with the school early teacher. A control group will consist of school implementing their usual teaching activities.

ELIGIBILITY:
Educational institutions that meet the following inclusion criteria will be invited to participate:

Inclusion Criteria:

1. Municipal or subsidized educational institutions.
2. Mixed educational institutions.
3. Educational institutions with preschool education with at least one class per level.
4. Educational institutions with a high vulnerability index, given by IVESINAE ≥ 75%.

Exclusion Criteria:

A criterion for exclusion will be educational institutions that are already developing or implementing a manualized program to promote social-emotional skills or participating in a similar study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 5 months
  Acceptability of the intervention will be assessed using qualitative questionnaires
Feasibility | 5 months
  Feasibility will be assessed by looking at the number of students successfully completing the study
Parental report of psychological difficulties | 8 months
  The psychological difficulties will be assessed using the total subscale of difficulties of the Parents version of The Strengths and Difficulties Questionnaire (SDQ)
Parental report of psychological strengths | 8 months
  The psychological strengths will be assessed using the total subscale of difficulties of the Parents version of The Strengths and Difficulties Questionnaire (SDQ)

SECONDARY OUTCOMES:
Teacher report of psychological difficulties | 8 months
  The psychological difficulties will be assessed using the total subscale of difficulties of the Teacher version of The Strengths and Difficulties Questionnaire (SDQ)
Teacher report of psychological strengths | 8 months
  The psychological strengths will be assessed using the total subscale of difficulties of the Teacher version of The Strengths and Difficulties Questionnaire (SDQ)
Executive function | 8 months
  Scores on the The Minnesota Executive Function Scale (MEFS)
Recognition of emotions | 8 months
  Scores on the Assessment of Children's Emotions Scale (ACES)
Social problem solving skills | 8 months
  Scores on the Challenging Situations Task (CST)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gaete, MD, MSc, PhD, Principal Investigator — Universidad de Los Andes; Marcelo Sanchez, MSc, Principal Investigator — Fundacion San Carlos de Maipo
Locations (1):
- Fundacion San Carlos de Maipo, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vicente B, Kohn R, Rioseco P, Saldivia S, Levav I, Torres S. Lifetime and 12-month prevalence of DSM-III-R disorders in the Chile psychiatric prevalence study. Am J Psychiatry. 2006 Aug;163(8):1362-70. doi: 10.1176/ajp.2006.163.8.1362. PMID 16877648
- [Background] Vicente B, Saldivia S, de la Barra F, Kohn R, Pihan R, Valdivia M, Rioseco P, Melipillan R. Prevalence of child and adolescent mental disorders in Chile: a community epidemiological study. J Child Psychol Psychiatry. 2012 Oct;53(10):1026-35. doi: 10.1111/j.1469-7610.2012.02566.x. Epub 2012 May 31. PMID 22646991
- [Background] Patel V, Chisholm D, Parikh R, Charlson FJ, Degenhardt L, Dua T, Ferrari AJ, Hyman S, Laxminarayan R, Levin C, Lund C, Medina Mora ME, Petersen I, Scott J, Shidhaye R, Vijayakumar L, Thornicroft G, Whiteford H; DCP MNS Author Group. Addressing the burden of mental, neurological, and substance use disorders: key messages from Disease Control Priorities, 3rd edition. Lancet. 2016 Apr 16;387(10028):1672-85. doi: 10.1016/S0140-6736(15)00390-6. Epub 2015 Oct 8. PMID 26454360
- [Background] Bould H, Araya R, Pearson RM, Stapinski L, Carnegie R, Joinson C. Association between early temperament and depression at 18 years. Depress Anxiety. 2014 Sep;31(9):729-36. doi: 10.1002/da.22294. Epub 2014 Aug 8. PMID 25111741
- [Background] Garber J, Clarke GN, Weersing VR, Beardslee WR, Brent DA, Gladstone TR, DeBar LL, Lynch FL, D'Angelo E, Hollon SD, Shamseddeen W, Iyengar S. Prevention of depression in at-risk adolescents: a randomized controlled trial. JAMA. 2009 Jun 3;301(21):2215-24. doi: 10.1001/jama.2009.788. PMID 19491183
- [Background] Domitrovich CE, Durlak JA, Staley KC, Weissberg RP. Social-Emotional Competence: An Essential Factor for Promoting Positive Adjustment and Reducing Risk in School Children. Child Dev. 2017 Mar;88(2):408-416. doi: 10.1111/cdev.12739. Epub 2017 Feb 18. PMID 28213889
- [Background] Denham SA. Social-Emotional Competence as Support for School Readiness: What Is It and How Do We Assess It? Early Education and Development, 17(1), 57-89, 2006.
- [Background] Garner PW, Waajid B. Emotion Knowledge and Self-Regulation as Predictors of Preschoolers' Cognitive Ability, Classroom Behavior, and Social Competence. Journal of Psychoeducational Assessment, 30(4), 330-343, 2012. doi:10.1177/0734282912449441
- [Background] Shure MB. I Can Problem Solve (ICPS). An interpersonal cognitive problem solving program (preschool). Champaign, IL: Research Press, 1992.
- [Background] Jones S, Brush K, Bailey R, Brion-Meisels G, McIntyre J, HKahn J, et al. Navigating SEL from the Inside Out. Looking inside and across 25 leading SEL programs: A practical resource for schools and OST providers. 2017.
- [Result] Shure MB, Spivack G. Interpersonal problem-solving in young children: a cognitive approach to prevention. Am J Community Psychol. 1982 Jun;10(3):341-56. doi: 10.1007/BF00896500. PMID 7113996
- [Result] Boyle D, Hassett-Walker C. Reducing Overt and Relational Aggression Among Young Children. Journal of School Violence, 7(1), 27-42, 2008. doi:10.1300/J202v07n01_03
- [Derived] Gaete J, Sanchez M, Nejaz L, Otegui M. Mental Health Prevention in Preschool Children: study protocol for a feasibility and acceptability randomised controlled trial of a culturally adapted version of the I Can Problem Solve (ICPS) Programme in Chile. Trials. 2019 Mar 4;20(1):158. doi: 10.1186/s13063-019-3245-3. PMID 30832708
- See also: Home page of Fundación San Carlos de Maipo — http://www.fsancarlos.cl
- See also: Home page of Universidad de los Andes — http://www.uandes.cl